CLINICAL TRIAL: NCT06676449
Title: Tumor Draining Lymph Nodes Sparing Radiotherapy Plus Immunotherapy and Chemotherapy in Locally Advanced Esophageal Squamous Cell Carcinoma: a Randomized Phase III Trial
Brief Title: TDLN-sparing RT Plus Immunotherapy and Chemotherapy in Locally Advanced ESCC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Kuai Le Zhao, MD, Prof., Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESO-Shanghai 26
Record Dates: First submitted 2024-11-05; First posted 2024-11-06 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Esophageal Carcinoma; Radiotherapy; Immunotherapy
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Immunotherapy; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Concurrent Immunotherapy plus TDLN-sparing RT and Chemotherapy (Experimental): PD-1 inhibitors will be administered intravenously, a fixed dose of 200 mg, once every 3 weeks for 1 year.
  Paclitaxel 135mg/m2 d1, cisplatin 25mg/m2 d1-3, once every 3 weeks for 4 cycles, or other guideline recommended regimens for 4 cycles.
  TDLN-sparing radiotherapy 50.4Gy/28Fx.
  Interventions: Drug: Immunotherapy; Drug: chemotherapy: Paclitaxel/Cisplatin or other guideline recommended regimens; Radiation: TDLN-sparing RT
- TDLN-sparing RT and Chemotherapy (Active Comparator): Paclitaxel 135mg/m2 d1, cisplatin 25mg/m2 d1-3, once every 3 weeks for 4 cycles, or other guideline recommended regimens for 4 cycles.
  TDLN-sparing radiotherapy 50.4Gy/28Fx. It is allowed to accept immunotherapy followed by radiotherapy.
  Interventions: Drug: chemotherapy: Paclitaxel/Cisplatin or other guideline recommended regimens; Radiation: TDLN-sparing RT

INTERVENTIONS:
Drug: Immunotherapy — PD-1 inhibitors will be administered intravenously, a fixed dose of 200 mg, once every 3 weeks for 1 year.
  Arms: Concurrent Immunotherapy plus TDLN-sparing RT and Chemotherapy
Drug: chemotherapy: Paclitaxel/Cisplatin or other guideline recommended regimens — Paclitaxel 135mg/m2 d1, cisplatin 25mg/m2 d1-3, once every 3 weeks for 4 cycles.
  or other guideline recommended regimens
Radiation: TDLN-sparing RT — TDLN-sparing radiotherapy 50.4Gy/28Fx.

SUMMARY:
The goal of this clinical trial is to learn if immunotherapy in combination with tumor draining lymph nodes-sparing radiotherapy (TDLN-sparing RT) and chemotherapy works to treat locally advanced esophageal squamous cell cancer in adults.

Researchers will compare immunotherapy in combination with TDLN-sparing RT and chemotherapy to TDLN-sparing RT and chemotherapy to see if immunotherapy works more effectively when using TDLN-sparing RT to treat locally advanced esophageal squamous cell cancer

Participants will:

TDLN-sparing RT for esophageal cancer 50.4Gy/28Fx Paclitaxel plus cisplatin every 3 weeks for 4 cycles PD-1 inhibitors or observation every 3 weeks for 1 year

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Aged 18-75 years
3. Histologically confirmed esophageal squamous cell carcinoma
4. Clinical stages T2-4N0M0 or TxN+M0 or TxNxM1 (Only for supraclavicular lymph nodes metastasis) based on the 8th UICC-TNM classification

7. Eastern Cooperative Oncology Group(ECOG) performance status: 0-1 8. Life expectancy ≥3 months 9. Adequate organ functions Absolute neutrophil counts (ANC) ≥1.5×109⁄L; Hemoglobin (Hb) ≥9g⁄dl; Platelet (Plt) ≥100×109⁄L; Total bilirubin ≤1.5 upper limit of normal (ULN); Aspartate transaminase (AST) ≤2.5 ULN; Alanine aminotransferase (ALT) ≤2.5 ULN; Creatinine ≤1.5 ULN 10.Received no more than 3 cycles immunotherapy and/or chemotherapy

Exclusion Criteria:

1. Esophageal perforation or hematemesis
2. Any active autoimmune disease or a history of autoimmune disease (such as the following, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism and hypothyroidism (effective hormone replacement therapy excepted)) and immunosuppressive agents or systemic hormonal therapy indicated within 28 days (for adverse events of chemoradiotherapy excepted).
3. Allergic to macromolecular protein preparations, or to any of the ingredients in PD-1 inhibitors for injection.
4. Uncontrolled heart diseases or clinical symptoms, such as: (1) New York Heart Association(NYHA) class II or higher heart failure; (2) unstable angina; (3) myocardial infarction within 1 year; (4)clinically significant arrhythmia requiring clinical intervention.
5. Congenital or acquired immunodeficiency (such as HIV infection); active hepatitis B (HBV-DNA≥104 copy number/ml) or hepatitis C (positive hepatitis C antibody, and HCV-RNA is higher than the detection limit of the analytical method); active tuberculosis.
6. Active infection or unexplained fever >38.5 °C within 2 weeks before randomization (fever due to tumor excepted, according to investigator).
7. Patients with fertility reluctant to take contraceptive measures during the trial, or female patients pregnant or breastfeeding.
8. According to the investigator, other factors that may cause termination of the study. ie, other serious diseases (including mental illness) require combined treatment, family or social factors, which may affect the safety or the collection of trial data.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2028-10-31 (Estimated); Study Completion 2030-10-30 (Estimated)

PRIMARY OUTCOMES:
PFS for patients with TDLN V15 ≤ 50% | 2 years
PFS for all patients | 2 years

SECONDARY OUTCOMES:
OS for patients with TDLN V15 ≤ 50% | 2 years
OS for all patients | 2 years
Adverse events | up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided